CLINICAL TRIAL: NCT01858597
Title: Endocrine Fibroblast Growth Factor 19 and 21 Regulate the Insulin Resistance State in Gestational Diabetes Mellitus
Brief Title: Fibroblast Growth Factors 19 and 21 in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Dongyu Wang, M.D., First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5010dong
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Results first posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM, FGF
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gestational diabetes mellitus (Other): Those women (subjects) with gestational diabetes mellitus
  Interventions: Diagnostic Test: biachemical detection
- control (Other): Those healthy pregnant women
  Interventions: Diagnostic Test: biachemical detection

INTERVENTIONS:
Diagnostic Test: biachemical detection — Serum FGF19 and FGF21 levels were determined by enzyme-linked immunosorbent assay (ELISA) and were correlated with anthropometric, metabolic, and endocrine parameters. Homeostasis model assessment (HOMA-IR) index was calculated and analysed.
  Second, samples for measurement were obtained from 30 women with GDM and 35 healthy pregnant controls undergoing caesarean sections at term. mRNA and protein expression levels of FGF19/FGF21 and their co-receptor βKlotho（KLB）in placenta, rectus muscle and subcutaneous fat tissues were investigated with real-time quantitative polymerase chain reaction (qRT-PCR), western-blot and immunohistochemistry (IHC), respectively. Clinical data were collected and analysed.

SUMMARY:
Gestational diabetes mellitus (GDM) is the most common complication in pregnancy. Both mother and offspring have a significantly increased future risk for metabolic and cardiovascular disease as a consequence of GDM. Pathological insulin resistance and the pancreatic β-cell dysfunction may contribute to the development and adverse outcomes of GDM.

Recently, fibroblast growth factor 19 (FGF19) and FGF21 have emerged as key endocrine regulators of glucose, lipid and energy metabolism. Both factors activate FGFRs in the context of co-receptor βKlotho(KLB) expression. After that, both proteins alter ERK phosphorylation and stimulate glucose uptake. Furthermore, these two factors ameliorate insulin resistance through various ways including up-regulating insulin mRNA, IRS-1, GLUT-1 expressions, down-regulating GH-IGF-1 levels in different tissues and blood circulation and also improving dyslipidemia.

Our previous studies showed that several factors which involved in insulin resistance and FGF19/FGF21 signaling pathway had differential expression in placenta from GDM and normal glucose tolerance pregnancy. Those led us to hypothesize that FGF19/FGF21 signaling pathway could play an important role in the pathogenesis and development of insulin resistance state in GDM.

In the present study, we will further investigate whether maternal and neonatal FGF19/FGF21 signaling pathway are altered and associated with insulin resistance, glucose intolerance, dyslipidemia and adverse pregnancy outcomes. Thus we will evaluate the regulating action of FGF19/FGF21 on gestational insulin resistance.

The aim of this study is to elucidate the role of FGF19/FGF21 in insulin resistance and metabolic disorder in GDM.

DETAILED DESCRIPTION:
First，30 pregnant women with GDM and 60 pregnant control women with normal glucose tolerance (NGT) matched for maternal and gestational age were enrolled in the study. All the subjects underwent antepartum screening in the First Affiliated Hospital of Sun Yat-sen University. Blood samples were obtained after overnight fasting at the time of oral glucose tolerance test (OGTT). Serum FGF19 and FGF21 levels were determined by enzyme-linked immunosorbent assay (ELISA) and were correlated with anthropometric, metabolic, and endocrine parameters. Homeostasis model assessment (HOMA-IR) index was calculated and analysed.

Second, samples for measurement were obtained from 30 women with GDM and 35 healthy pregnant controls undergoing caesarean sections at term. mRNA and protein expression levels of FGF19/FGF21 and their co-receptor βKlotho（KLB）in placenta, rectus muscle and subcutaneous fat tissues were investigated with real-time quantitative polymerase chain reaction (qRT-PCR), western-blot and immunohistochemistry (IHC), respectively. Clinical data were collected and analysed.

Data were analyzed by SPSS 20.0 database. The results were expressed as mean ± standard deviations or median with interquartile range. Differences between groups were assessed by Student's unpaired t test, Mann-Whitney U test, or Chi-square test as appropriate. Correlation analysis was performed using the Spearman rank correlation method. To identify independent relationships and adjust the effects of covariates, multiple linear regression analyses were performed. P values of <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy;
* Regular antenatal examination from the first trimester;
* Give birth in the university hospital (The 1st affiliated hospital of Sun Yat-sen University)

Exclusion Criteria:

* Younger than 18 years old;
* Older than 40 years old;
* Multiple pregnancy;
* Diagnosed DM before pregnancy;
* Complicated with other diseases such as hypertension, eclampsia, thyroid diseases, etc.;
* Taking any drug that affect glucose and lipid metabolism and insulin sensitivity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zilian Wang, M.D., PhD, Study Director — Obstetrics and Gynechology Department of the 1st affiliated hospital of SYSU
Locations (1):
- Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Gestational Diabetes Mellitus: Women with gestational diabetes mellitus.
- Control: Women with normal glucose tolerance.
Period: Overall Study
Arm/Group | Gestational Diabetes Mellitus | Control
Started | 30 | 60
Completed | 30 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gestational Diabetes Mellitus: Women with gestational diabetes.
- Total: Total of all reporting groups
Arm/Group | Gestational Diabetes Mellitus | Control | Total
Number analyzed (Participants) | 30 | 60 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 60 | 90
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 60 | 90
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 60 | 90

OUTCOME MEASURES:

1. Primary Outcome: The Concentration of Serum FGF19
Time Frame: in fasting state during 24-28 gestational weeks
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Gestational Diabetes Mellitus | Control
Number analyzed (Participants) | 30 | 60
pg/mL | 65.96 [51.76 to 90.11] | 124.47 [82.72 to 189.50]

2. Secondary Outcome: Expression of FGF19 in Term Placenta
Time Frame: term delivery (when participants come back to hospital to give birth during 37-41 gestational weeks)
Population: In this study we included 90 cases with serum samples as well as 45 term deliveries with placenta samples. The secondary outcome was to analyze the expression of FGF19 in term placenta, therefore only 45 cases were included.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Gestational Diabetes Mellitus | Control
Number analyzed (Participants) | 20 | 25
pg/mL | 0.33 (0.05) | 0.72 (0.09)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 10 months
Description: There are no adverse events in this study.
Arm/Group | Gestational Diabetes Mellitus | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/60
Other Adverse Events (participants affected / at risk) | 0/30 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes